CLINICAL TRIAL: NCT04440449
Title: Effect of Behavioral Lifestyle Intervention on Frailty in Older Adults With Diabetes: A Pilot Study
Brief Title: Effect of Behavioral Lifestyle Intervention on Frailty in Older Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rozmin Jiwani, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20190019H; P30AG044271 (NIH)
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Frailty; Weight, Body; Type 2 Diabetes
MeSH Terms: conditions — Frailty; Body Weight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: * Group A - Mobile Health + group intervention
  * Group B (control arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Lifestyle Intervention (Experimental): The participants will receive behavioral lifestyle intervention with a smartphone-based self-monitoring for diet and physical activity. This group also includes a total of 10 Group sessions over 6 months.
  Interventions: Behavioral: Lifestyle App; Behavioral: Look AHEAD behavior lifestyle intervention
- Group B control arm (Other): Participants use the smart-phone app to record their daily diet and physical activity, with no group sessions.
  Interventions: Behavioral: Lifestyle App; Behavioral: Abbreviated Look AHEAD behavior lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle App — A mobile app used to assist with lifestyle changes
Behavioral: Look AHEAD behavior lifestyle intervention — A modified Look AHEAD behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity
  Arms: Behavioral Lifestyle Intervention
Behavioral: Abbreviated Look AHEAD behavior lifestyle intervention — An abbreviated Look AHEAD behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity
  Arms: Group B control arm

SUMMARY:
The study team want to see if changes in lifestyle and behaviors and self-monitoring of diet and physical activity in older adults who have type 2 Diabetes (T2D) may help to prevent or reduce frailty. Frailty occurs in older adults and leads people to have falls, become disabled, require nursing home placement, and have increased risk of death. T2D is one of the major risk factors for frailty. T2D is a significant problem in older adults and is known to increase the risk of future frailty.

DETAILED DESCRIPTION:
Behavioral lifestyle intervention: Participants (N=40) will be randomized to the mHealth+ group Intervention group (Group A; n=20)and mHealth+ individual intervention group (Group B; n=20) group using a randomization table. (1) The mHealth+ group Intervention group (Group A) will receive a modified Look AHEAD behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity. This comprises ten group sessions for lifestyle intervention in 6-months. The group will receive three weekly classes in the first month and then bi-weekly classes for month 2-3, and three monthly session in month four, five, and six. The frequency and layout of these classes will allow participants to master new skills gradually, then eventually wean off, and adopt the modified lifestyle as the part of their daily lives. (2) The mHealth+ individual intervention group (Group B) will receive an abbreviated behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity in one face-to-face individual session at the beginning of the study. In addition, participants will receive self-study materials, from Look Ahead modules, and a monthly follow-up phone calls for the duration of the study (6-months). The goal for these follow up phone calls are to assess understanding of the modules, to promote continued engagement with the study material, and to provide clarification on materials as needed. Participants in the mHealth+ group Intervention group (Group A) and mHealth+ individual intervention group (Group B will receive instruction on how to download an app to help them record their diet and physical activity at the beginning of the study.

Fitbit offers a simple, easy-to-use tool for tracking food and physical activity. It helps set daily calorie budget, and set and work towards goals for nutrient intake, weight loss, exercise, and more. https://www.fitbit.com/inspire 04.12.20: Due to SARS-CoV2 (COVID-19) and social distancing order, the study team are adding hemoglobin Hba1c home test.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Age 65 and older
* Men and women of all ethnic groups
* Self-reported of provider-diagnosed with Type 2 Diabetes (T2D) for at-least 6 months.
* Received basic diabetes self-management education
* Stable medication regimen and no medication changes are expected over the next 6 months.
* Overweight/obese (Body Mass Index (BMI) ≥25 kg/m2
* Able to read and write in English
* Own a smartphone
* At PI discretion, participant is willing/able to comply with the protocol requirements

Exclusion Criteria:

* Unsafe to walk using Exercise Assessment and Screening for You (EASY) criteria or clinical judgement of the PI.
* History of severe psychiatric disorders or cognitive impairment which interferes with active participation in the study
* Residence of long-term care facility
* History of substance abuse in the past year
* Unwilling to be randomized in a Mobile Health (mHealth+) individual intervention group

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozmin Jiwani, RN, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared with mentors and advisors
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available at study completion
Access Criteria: Study Teams plans on publication at completion of data analysis.

REFERENCES:
- See also: J. Frailty Aging 2021 April 24: 1-9 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8068458/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The control group did not recruit any subjects due to the COVID-19 pandemic
Groups:
- Behavioral Lifestyle Intervention: This group will receive behavioral lifestyle intervention with a smartphone-based self-monitoring for diet and physical activity. This group also includes a total of 10 Group sessions over 6 months.
  Lifestyle App: A mobile app used to assist with lifestyle changes
- Group B - Control Group: The mHealth+ individual intervention group (Group B) will receive an abbreviated behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity in one face-to-face individual session at the beginning of the study. In addition, participants will receive self-study materials, from Look Ahead modules, and a monthly follow-up phone calls for the duration of the study (6-months)
Period: Overall Study
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group
Started | 20 | 0
Completed | 18 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants were older adults with Type 2 diabetes. Group B did not enroll any participant due to the COVID-19 pandemic.
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group | Total
Number analyzed (Participants) | 18 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (5.3) |  | 71.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 |  | 10
  Male | 8 |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 |  | 9
  Not Hispanic or Latino | 9 |  | 9
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 |  | 18

OUTCOME MEASURES:

1. Primary Outcome: Frailty Scale Using Fried's Phenotype Method Based on Five Frailty Characteristics
Description: 1. Self-reported (SR) exhaustion (Y/N ) on Center for Epidemiologic Studies Depression (CES-D) scale: "Do you feel full of energy?" "No" scored a 1 (exhausted).
  2. SR unintentional weight loss: "In the last year, have you lost more than 10 pounds unintentionally?". "Yes" scored a 1.
  3. SR physical activity over the last year using the Minnesota Leisure Time Activity Questionnaire, (energy expenditure in kcal/week, standardized for sex). The lowest quintile for each sex group received a score of 1
  4. Grip strength measured (Kg) with a dynamometer in the dominant hand, standardized using body mass index quartiles and sex. The average of 3 trials was recorded. The lowest quintile for each sex group received a score of 1 (for weak).
  5. 10 feet walked at usual pace, standardized based on height and sex. The fastest of 2 trials was recorded. Participants in the lowest quintile for each sex group were considered slow (score =1) A higher scale score from 0-5 indicates greater frailty
Time Frame: Baseline to 6 months
Population: The control group did not recruit any subjects due to the COVID-19 pandemic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group
Number analyzed (Participants) | 18 | 0
score on a scale
  Baseline | 1.61 (1.15) |
  6 months | 0.94 (0.94) |
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention; Test type: Superiority; p = 0.01, t-test, 2 sided

2. Secondary Outcome: Glycated Hemoglobin (HbA1c)
Description: Change in HbA1c measured over the study period
Time Frame: Baseline to 6 months
Population: The control group did not recruit any subjects due to the pandemic
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin
Groups:
- Group B -Control Group: The mHealth+ individual intervention group (Group B) will receive an abbreviated behavior lifestyle intervention with smartphone-based self-monitoring of diet and physical activity in one face-to-face individual session at the beginning of the study. In addition, participants will receive self-study materials, from Look Ahead modules, and a monthly follow-up phone calls for the duration of the study (6-months)
Arm/Group | Behavioral Lifestyle Intervention | Group B -Control Group
Number analyzed (Participants) | 18 | 0
Percentage of glycated hemoglobin
  Baseline | 6.95 (0.84) |
  6 months | 6.75 (0.95) |
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention; Test type: Superiority; p = 0.108, t-test, 2 sided

3. Secondary Outcome: Short Physical Performance Battery (SPPB) Balance
Description: The balance test assesses a person's ability to stand with the feet together in side-by-side, semi-tandem, and full-tandem positions for 10 seconds each, responses ranging between 0-4 with a higher score indicating better balance. Three balance tests are performed and scoring is as follows:
  Side-by-side stand: person attempts to stand with feet together, side-by-side, for 10 seconds.
  * 1 point if held for 10 seconds
  * 0 points if not held for 10 seconds or not attempted Semi-tandem stand: person attempts to stand with the side of the heel of one foot touching the big toe of the other foot for 10 seconds.
  * 1 point if held for 10 seconds
  * 0 points if not held for 10 seconds or not attempted Tandem stand: person attempts to stand with the heel of one foot in front of and touching the toes of the other foot for about 10 seconds.
  * 2 points if held for 10 seconds
  * 1 point if held for 3 to 9.99 seconds
  * 0 points if held for <3 seconds or not attempted
Time Frame: Baseline to 6 months
Population: The control group did not recruit any subjects due to the COVID-19 pandemic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group
Number analyzed (Participants) | 18 | 0
score on a scale
  Baseline | 3.39 (0.78) |
  6 months | 3.89 (0.47) |

4. Secondary Outcome: SPPB Gait Speed
Description: Gait speed at a 4-meter walk is timed in seconds as participants walk at their usual pace. Two trials were administered, time (in seconds) was recorded for each trial. The fastest walk of two trials was recorded. Score is recorded between 0-4 with a higher score indicating a faster gait speed. Scoring is as follows:
  * 0 points if unable to do the walk
  * 1 point if time is more than 8.70 sec
  * 2 points if time is 6.21 to 8.70 sec
  * 3 points if time is 4.82 to 6.20 sec
  * 4 points if time is less than 4.82 sec
Time Frame: Baseline to 6 months
Population: Group B did not recruit any subjects due to the COVID-19 pandemic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group
Number analyzed (Participants) | 18 | 0
score on a scale
  Baseline | 3.61 (0.61) |
  6 months | 3.72 (0.57) |

5. Secondary Outcome: SPPB Chair Stands
Description: Chair stand represents the time to complete five chair rises, sit to stand from a chair, as quickly as possible, without using hands, responses ranging between 0-4. Scoring is as follows:
  * 0 points if unable to complete 5 chair stands or completes stands in >60 seconds
  * 1 point if chair stand time is 16.70 sec or more
  * 2 points if chair stand time is 13.70 to 16.69 sec or more
  * 3 points if chair stand time is 11.20 to 13.69 sec
  * 4 points if chair stand time is 11.19 sec or less
Time Frame: Baseline to 6 months
Population: Group B did not recruit any subjects due to the COVID-19 pandemic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Group B - Control Group
Number analyzed (Participants) | 18 | 0
score on a scale
  Baseline | 2.28 (1.27) |
  6 months | 2.44 (1.04) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected during active study participation, from baseline to 6 months
Arm/Group | Behavioral Lifestyle Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04440449/Prot_SAP_000.pdf